CLINICAL TRIAL: NCT05217199
Title: The Prechtl's General Movement Assessment, Hammersmith Infant Neurological Examination and Sensory Profile-2 in Prediction of Cerebral Palsy at Two Years of Age in High-Risk Infants: A Retrospective Study
Brief Title: The Prechtl's General Movement Assessment, Hammersmith Infant Neurological Examination and Sensory Profile-2
Acronym: highrisk
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, Assistant Proffessor, Kahramanmaras Sutcu Imam University
Other Study IDs: KSU3
Record Dates: First submitted 2022-01-05; First posted 2022-02-01 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Infant Development; Sensory Disorder; Sensory Processing Disorder; Motor Delay; Infant, Premature, Diseases; Infant, Very Low Birth Weight; Infant Asphyxia; Development Delay
Keywords: Motor development; Sensory development; High risk of Infants; Sensry disorder
MeSH Terms: conditions — Sensation Disorders; Psychomotor Disorders; Infant, Premature, Diseases; Learning Disabilities | interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/high risk of infants for cp: 1/ high risk of infants for cp was evaulated.
  Interventions: Other: Measurements

INTERVENTIONS:
Other: Measurements — Demographic information of infants and parents, prenatal, postnatal and natal risk factors, Magnetic Resonance Images (MRI), General Movements (GMs) evaluations of babies with Prechtl method from NICU will be recorded. Video recordings for General Movements (GMs) analyzes with the Prechtl method will be taken at postterm 12th to 20th weeks. The infants' sensory processing (general, auditory, visual, tactile, movement, oral) will be evaluated with the adjusted Infant Sensory Profile-2 (ISP-2) family scale, which will be filled in by their mothers at the 3rd month. For motor assessments, the postterm corrected 3 month Hammersmith Infant Neurological Examination (HINE) will be used. A pediatric neurologist who was blinded to all testing made the diagnosis of CP in a 2-year-old child based on neuroimaging and clinical tests.

SUMMARY:
In the Neonatal Intensive Care Unit (NICU), infants encounter many sensory stimuli (excessive noise, bright lights, painful medical applications, etc.) that are not present in the uterus. During the critical period of brain development, this sensory overload affects the physiological responses of infants; It can lead to sensory processing problems by causing negative changes in motor, neurological and sensory development. Sensory processing was explained by Dunn as the emergence of appropriate reactions and behaviors in neurological processes in which visual, auditory, tactile, oral, olfactory, vestibular, proprioceptive and kinesthetic inputs are regulated.

DETAILED DESCRIPTION:
There are interactions between an individual's neurological thresholds and emotional and behavioral responses or self-regulation strategies. Sensory modulation is an active processing process in which the brain adapts to sensory inputs from the environment by stimulating or inhibiting neurons as required by the current situation. Based on the interaction between an individual's neurological threshold and behavioral responses, Dunn developed four different response categories. These are sensation seeking, avoidance, low registration, and increased sensory sensitivity. From infancy, these processes show appropriate development with natural stimuli. However, sometimes there may be deviations in development from early infancy. One of them is the NICU, which is necessary to support vital functions. Decreased spontaneous movements for any reason and exposure to excessive sensory stimuli in this environment may cause negative consequences for the normal sensory and motor development of the baby.Babies who stay in the NICU for a long time stay away from natural sensory stimuli. Newborn preterm infants receive less tactile and vestibular stimulation in the NICU than does prenatal maternal movement. However, they are exposed to increased stimulus with other negative stimuli such as bright lights, high noise levels, excessive use and frequent painful interventions, which are not found in the intrauterine environment in the NICU. This can have lasting effects on the developing brain and affect the natural development of sensory systems. In the studies conducted, a significant difference was found between term babies and preterm babies in terms of sensory profile scores. Studies examining the relationship between sensory processing parameters and motor development in infants are limited in the literature. There is also a need for studies examining the relationship between sensory-motor development from the neonatal period. It is thought that preterm infants are exposed to these negative sensory stimuli longer. Neurodevelopmental follow-up is required after discharge in these infants with biological sensitivity and risk of neurological injury.The aim of this study is to examine the motor and sensory development of high-risk infants and compare them with their peers.

ELIGIBILITY:
Inclusion Criteria:

* Term preterm babies with 0-3 months of prenatal, postnatal and natal risk who stayed in the NICU for >2 weeks for any reason and were corrected after discharge
* Babies with periventricular bleeding, ICH stage 2, 3, 4, cystic PVL, stage 3 HIE, neonatal bilirubin encephalopathy (kernicterius), perinatal stroke, perinatal asphyxia, hydrocephalus
* Babies with chronic lung disease, RDS, BPD and long-term Oxygen support (≥7 days)
* Preterm infants with gram-negative bacteria-associated sepsis, Necrotizing Enterocolitis (NEC), infantile apnea, cerebral malformation
* Preterm babies with low 5th minute Apgar score (3 and below), diagnosed with intrauterine growth retardation, multiple births (twins, triplets), PR
* Infants with prolonged severe hypoglycemia and hypocalcemia
* Surgical conditions such as diaphragmatic hernia or tracheoesophageal fistula
* Babies who are small for gestational age (GYB, less than 3rd percentile) or large for gestational age (GYB, greater than 97th percentile)
* Babies who are MV dependent for more than 24 hours
* Babies born less than 32 weeks of gestation and weighing less than 1500 g
* Healthy term babies

Exclusion Criteria:

* - Babies of parents who did not agree to participate in the study/Babies who did not attend follow-up evaluations
* Babies with congenital malformations (Spina Bifida, Congenital Muscular Torticollis, Arthrogryposis Multiplex Congenita)
* Babies diagnosed with metabolic and genetic diseases (Down Syndrome, Spinal Muscular Atrophy, Duchenne Muscular Dystrophy.)
* Babies who are still intubated and dependent on MV at postterm 3 months
* Babies with hearing and vision loss

Ages: 25 Weeks to 42 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: High risk of infants and healty peer aged control group
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Infant Sensory Profile-2 (ISP-2) | one assessment at the corrected age of 3th months.
  The Infant Sensory Profile (ISP-2) questionnaire is a 24-item questionnaire consisting of sensory profile general sensory processing score, auditory processing, visual processing score, tactile processing, motion processing, oral sensory processing sub-scores. The sensory profile raw score total score is calculated with the sum of the sub-scores. Higher scores shows better sensory functions.
Hammersmith Infant Neurological Examination (HINE) | one assessment at postterm corrected age of 3th months.
  The HINE is a simple, standardized, and scorable test for the clinical neurological evaluation of 2-to-24-month-old infants. It has 3 sections: (1) neurological examination (26 items, scored) evaluating cranial nerve function, posture, movements, tone, reflexes, and reactions, (2) motor milestones (8 items, unscored), and (3) behaviour (3 items, unscored). Each of the 26 items is scored first separately (as 0, 1, 2, or 3, half scores) and then the total score is calculated with a maximum score of 78. Higher score indicates good neurological function.
Prechtl's General Movements Assessments (GMs)1 | Measurement at postterm age of 12tk to 20th weeks.
  General movements (GMs) are the spontaneous movement repertoire present from early foetal life until 20 weeks post-term. From birth to 8 post-term weeks, they have a "writhing" character. They will be scored as cs-pr-n-ch. From 12th to 20th weeks, they have "fidgety" character.
Diagnosis of CP (neuroimaging by MRI) | Measurement once at 2 years of age
  Based on neuroimaging and clinical evaluations at 2 years of age, a pediatric neurologist who was blinded to all assessments diagnosed CP. The neuroimaging scans were classified into one of seven primary patterns of abnormality as defined and described by

CONTACTS AND LOCATIONS:
Overall Officials: hatice adıgüzel, PhD, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Hatice Adıgüzel, Kahramanmaraş, Dulkadiroglu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No